CLINICAL TRIAL: NCT06082557
Title: A Clinical Study on the Observation and Evaluation on the Safety and Efficacy of T60c Injection in the Treatment of Patients With Advanced Solid Tumors
Brief Title: A Study to Observe and Evaluate the Safety and Efficacy of T60c Injection for Treatment of Advanced Solid Tumor Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, BING HE XU, Chief physician of Department of Medical Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T60c-017-2023
Record Dates: First submitted 2023-09-22; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Malignant Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All the subjects enrolled will receive the experimental intervention, T60c injection (Experimental)
  Interventions: Drug: T60c injection

INTERVENTIONS:
Drug: T60c injection — Peripheral blood mononuclear cells (PBMCs) are used for cell preparation. PD-1 positive T cells are isolated from peripheral blood by blood cell apheresis method and transduced with lentivirus loaded with "enhanced receptor" and "TROP2-CAR" (TROP2-chimeric antigen receptor). The obtained T60c is used for one-time intravenous infusion.

SUMMARY:
This is an open-labeled, single-arm, multiple-dose escalation and single-dose expansion clinical study of cell therapy to observe and evaluate the safety and efficacy of T60c injection in the treatment of patients with advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤80 years old, gender is not limited;
2. Life expectancy>3 months;
3. The Eastern Oncology Consortium (ECOG) performance status from 0 to 1;
4. Subjects with malignant solid tumors confirmed by pathological diagnosis（who have failed or unable to tolerate in standard treatment(s), or haven't received standard treatment），including：

   1. Breast cancer: including hormone receptor positive and triple negative breast cancer;
   2. Non-small cell lung cancer, digestive system tumors (esophageal cancer, gastric cancer, colorectal cancer, pancreatic cancer), urinary system tumors (urothelial cancer, prostate cancer), gynecological tumors (cervical cancer, endometrial cancer, ovarian cancer). And the TROP-2 expression rate of tumor tissue in IHC (immuno-histochemistry) staining is ≥ 50%.
5. The percentage of PD-1positive T lymphocytes in total T lymphocytes is more than 10%, and subjects should voluntarily receive peripheral blood mononuclear cell (PBMCs) apheresis collection.
6. At least one or more measurable lesions (CT slice thickness ≤ 5 mm, maximal diameter ≥ 10 mm, and lymph node with malignant metastasis minimal diameter of ≥15 mm) according by RECIST 1.1.
7. No serious hematological, hepatic, and renal function abnormalities, adequate function defined as :

   1. Blood system (no blood transfusion or hematopoietic stimulating factor treatment within 14 days): Neutrophil count (ANC) ≥1.5×109/L, Platelet (PLT) ≥75×109/L, Hemoglobin (Hb) ≥80g/L, Lymphocyte count (LYM) ≥ 60%×lower limit of normal value;
   2. Hepatic function: Total bilirubin (TBIL) ≤1.5×ULN, Alanine aminotransferase (ALT) ≤2.5×ULN,, Aspartate aminotransferase (AST) ≤5×ULN of patients with liver metastasis, Creatinine ≤1.5×ULN or creatinine clearance (eGFR) ≥60 mL/min (Cockcroft and Gault formula);
   3. Blood coagulation function: Activated partial thrombin time (APTT) ≤1.5×ULN, International normalized ratio (INR) ≤1.5×ULN;
8. Eligible subjects (male or female) must comply with effective contraception methods (hormonal or barrier method or abstinence, etc.) during the trial period at least 90 days after T60c injection treatment; Female subjects of childbearing potential (definition refers to appendix) must undergo a pregnancy test (blood or urine) and the results must be negative within 7 days prior to first use of T60c injection.
9. Subjects must be able to understand the protocol and be willing to enroll the study, sign the informed consent, and be able to comply with the study and follow-up procedures.

Exclusion Criteria:

1. Subjects with symptomatic and/or untreated brain metastases (of any size and number); However, subjects may be eligible if they received documented treatment, and the intracranial lesion(s) remain stable for at least 2 months before starting screening;
2. Subjects suffered from other malignant tumors within two years prior screen or concurrent malignancy, except for basal cell skin cancer that has been cured, and in situ malignancies of cervical carcinoma or lung cancer;
3. Subjects received treatment with tislelizumab (excluding other PD-1 monoclonal antibodies) or any PD-L1 monoclonal antibody within the first 12 weeks of screening;
4. Subjects received systemic chemotherapy, radiotherapy, immunotherapy and targeted therapy within 2 weeks before screening; However, the restriction for Nitroso urea or Mitomycin C are within 6 weeks before screening;
5. Subjects received chronic systemic sex hormone treatment for any reason within 12 weeks before screening; However, the use of low-dose glucocorticoid replacement therapy due to adrenal cortex dysfunction is exempted.
6. Subjects received granulocyte Colony-stimulating factor (G-CSF) and Granulocyte-macrophage colony-stimulating factor (GM-CSF) for leukocytosis within 12 weeks before screening;
7. Subjects received with Trop-2-targeted drug treatment previously;
8. Any active autoimmune disease or autoimmune disease in history, which is included but not limited to: autoimmune hepatitis, interstitial pneumonia, enteritis, vasculitis, nephritis; and asthma requiring medical intervention by bronchiectasis, etc., except for vitiligo, psoriasis and alopecia without systemic treatment, well controlled type I diabetes, hypothyroidism with normal thyroid function after replacement therapy;
9. Recipients of any organ transplant, including allogeneic stem cell transplants, with exception of transplants requiring no immunosuppression (e.g., corneal transplants, hair transplants);
10. Subjects with any forms of primary immunodeficiency (e.g., severe combined immunodeficiency disease (SCID) and acquired immunodeficiency syndrome (AIDS);
11. Presence of major acute or chronic infections, including:

    1. Viral hepatitis, including hepatitis B (HBsAg positive and/or hepatitis B DNA copy number higher than the lower detection threshold of the research center), Hepatitis C, etc.; HIV antibody test positive; Patients with positive Treponema pallidum antibodies;
    2. Active bacterial or fungal infections that require systemic treatment;
    3. Active tuberculosis infection with clinical symptoms, physical examination or imaging, and laboratory findings;
12. Acute exacerbation of chronic obstructive pulmonary disease or other respiratory diseases;
13. Cardiovascular/Cerebrovascular disease with clinical significance, such as cerebrovascular accident/stroke (<6 months before enrollment), myocardial infarction (<6 months before enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Class II) or severe arrhythmia;
14. Clinically uncontrollable serious cavity effusion which is judged by researchers as unsuitable for inclusion;
15. Subjects received any genetically modified cell therapy in the past;
16. Subjects need anticoagulant treatment (Warfarin or heparin);
17. Subjects need long-term antiplatelet therapy (including but not limited to: aspirin >300mg/d or clopidogrel >75mg/d, etc.);
18. Pregnant or lactating women;
19. Subjects with no/limited capacity for civil conduction, or mental disorders/ poor compliance;
20. Alcoholic or drug abuse;
21. Subjects or its families are incapable to understand the content and objectives of this clinical study;
22. Subjects with other serious or uncontrolled systemic diseases, or other conditions deemed unsuitable for participation in this clinical trial as judged by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate（ORR） | 3 months after T60c transfusion
  The number of cases with CR (complete remission) and PR (partial remission) accounted for the total number of evaluable cases
Disease Control Rate(DCR) | 3 months after T60c transfusion
  The number of cases with remission and stable lesions after treatment accounted for the total number of evaluable cases

SECONDARY OUTCOMES:
Progression-Free Survival(PFS) | From the day of T60c transfusion until the day of first documented progression or death from any cause, whichever came first, assessed up to 27 months.
  A time quantum from the day which subject received T60c transfusion to the day which subject was evaluated of the first disease progression or death due to any reasons.
Objective Response Rate（ORR） | through study completion, an average of 27 months.
  The number of cases with remission and stable lesions after treatment accounted for the total number of evaluable cases.
Duration of Response（DOR） | From the day that the subject was first evaluated as CR or PR to the day which subject was evaluated as PD or death due to any reasons, assessed up to 27 months.
  A time quantum from the day which subject first evaluated as CR or PR to the day which subject was evaluated as PD (progressive disease) or death due to any reasons.
Overall survival(OS) | From the day of T60c transfusion until the day of T60c transfusion to death due to disease, assessed up to 27 months.
  A time quantum from the day subject received T60c transfusion to death due to disease.

IPD SHARING:
Plan to Share IPD: No